CLINICAL TRIAL: NCT06314685
Title: A Single-center, Randomized, Blind, Positive Control Phase III Clinical Trial to Evaluate Immunogenicity and Safety of Group ACYW135 Meningococcal Polysaccharide Conjugate Vaccine in Healthy Volunteers Aged From 6 Months to 5 Years
Brief Title: Immunogenicity and Safety of MCV4 in Volunteers Aged 6 Months-5 Years
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2020040C-2
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-02

CONDITIONS: Healthy Population
Keywords: Group ACYW135 Meningococcal Polysaccharide Conjugate Vaccine; MCV4

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 6~11 months old (Experimental): For children aged 6-11 months, they was randomly assigned in a 1:1 ratio to the experimental group and control group, and basic immunization was performed following a 0,1-month schedule. And the experimental group received one dose of booster immunization at 18 months old;
  Interventions: Biological: Group ACYW135 Meningococcal Polysaccharide Conjugate Vaccine; Biological: Group A and C Meningococcal Polysaccharide Vaccine
- 12~23 months old (Experimental): For infants aged 12-23 months, they was randomly assigned in a 1:1:1 ratio to the two-dose experimental group, one-dose experimental group, and two-dose control group. For the 12-23 month-olds in the two-dose group, they received two doses of immunization according to a 0, 1-month schedule; while those in the one-dose group receive a single dose of immunization.
  Interventions: Biological: Group ACYW135 Meningococcal Polysaccharide Conjugate Vaccine; Biological: Group A and C Meningococcal Polysaccharide Vaccine
- 2~5 years old (Experimental): For children aged 2-5 years, they were randomly assigned in a 1:1 ratio to the experimental group and control group and received a single dose of immunization.
  Interventions: Biological: Group ACYW135 Meningococcal Polysaccharide Conjugate Vaccine; Biological: Group ACYW135 Meningococcal Polysaccharide Vaccine

INTERVENTIONS:
Biological: Group ACYW135 Meningococcal Polysaccharide Conjugate Vaccine — As a experimental vaccine for 6 months to 5 years old.
Biological: Group A and C Meningococcal Polysaccharide Vaccine — As a control vaccine for ages 6-11 months and 12-23 months.
  Arms: 12~23 months old; 6~11 months old
Biological: Group ACYW135 Meningococcal Polysaccharide Vaccine — As a control vaccine for ages 2-5 years.
  Arms: 2~5 years old

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of Group ACYW135 Meningococcal Polysaccharide Conjugate Vaccine in healthy volunteers aged from 3 months to 5 years old.

DETAILED DESCRIPTION:
This is a Phase III, single center, randomized, blind, positive control clinical trial conducted in Hunan Province, China. The purpose of this study is to evaluate the immunogenicity and safety of Group ACYW135 Meningococcal Polysaccharide Conjugate Vaccine in healthy volunteers aged from 3 months to 5 years old. A total of 2450 subjects were included, divided into three age groups: 6-11 months old (700 subjects), 12-23 months old (1050 subjects), and 2-5 years old (700 subjects).

ELIGIBILITY:
Inclusion Criteria:

For primary immunization stage:

* Subjects aged 6 months-5 years;
* Subjects should be full-term (37-42 weeks of gestation) and their birth weight should meet the requirements (2500g ≤ body weight ≤ 4000g);
* Axillary body temperature ≤ 37.0 ℃;
* The guardian of the subject voluntarily agrees to the child's participation in the study and signs an informed consent form;
* The guardians of the subjects have the ability to understand the research procedures and participate in all planned follow-up visits;
* Infants and young children aged 6 to 23 months have not received the meningococcal conjugate vaccine. If they have been vaccinated with group A meningococcal polysaccharide vaccine, the interval between vaccination and the previous dose should exceed 3 months;
* Children aged 2-5 who have not been vaccinated with meningococcal conjugate vaccine, if they have been vaccinated with meningococcal polysaccharide vaccine (including group A meningococcal polysaccharide vaccine, group A and C meningococcal polysaccharide vaccine, and group ACYW135 meningococcal polysaccharide vaccine), the interval between the last dose should exceed 12 months;
* Subjects had no vaccination history of other live attenuated vaccines (such as BCG vaccine, live attenuated polio vaccine, rotavirus vaccine, etc.) within 14 days before vaccination, and no vaccination history of other non live vaccines (such as hepatitis B vaccine, inactivated polio vaccine, DPT vaccine, etc.) within 7 days.
* Subjects who have not been vaccinated with meningococcal group A and C conjugate vaccine at the aged of 3-5 months;
* Subjects who had no history of other live vaccines within 14 days before vaccination and no history of other inactivated vaccines within 7 days;

For booster immunization stage (applicable to the 6-11 month age group):

* Infants and young children who have been enrolled in this clinical trial between 6 and 11 months of age and have reached the age of 18 months;
* Infants and young children who have completed basic immunization in this clinical trial;
* According to the opinions of the researchers, the subjects and their guardians are able to comply with the requirements of the clinical trial protocol.

For immune persistence stage (applicable to the 12-23 month age group):

* Children who have been enrolled in this clinical trial at 12-23 months of age and have completed basic immunization for 12 months; According to the researcher's opinion, the subjects and their guardians are able to comply with the requirements of the clinical trial protocol.

Exclusion Criteria:

For primary immunization stage:

* Have a history of severe allergic reactions that require medical intervention; Have a history of allergies to vaccines or vaccine ingredients (such as lactose, sodium chloride, tetanus toxoids, etc.), and other serious adverse reactions to vaccines;
* Has contraindications for intramuscular injection such as thrombocytopenia, any coagulation dysfunction, or undergoing anticoagulant therapy;
* Has severely abnormal labor (dystocia, instrumental delivery, excluding cesarean section), or history of asphyxia, neurological damage, in vitro fertilization or multiple pregnancy, pathological jaundice (only applicable to infants and young children aged 6-11 months);
* Suffering from serious congenital malformations or chronic diseases that may interfere with the progress or completion of the study (including but not limited to Down's syndrome, thalassemia (the first degree relatives in the family are thalassemia or gene carriers of thalassemia), heart disease, kidney disease, diabetes, autoimmune diseases (repeated perianal abscesses), hereditary allergies, Guillain Barre syndrome, etc.);
* Infectious diseases with clinical or serological evidence, such as tuberculosis, hepatitis B, hepatitis C, human immunodeficiency virus (HIV) infection or HIV infected parents;
* Any situation resulting in splenomegaly, splenectomy, or functional splenomegaly;
* Has a history of convulsions, epilepsy, encephalopathy, and mental illness (including family history);
* Within 3 days prior to the first dose of the vaccine, there was an acute illness or acute exacerbation of a chronic disease, or the use of antipyretic, analgesic, and anti allergic drugs (such as acetaminophen, ibuprofen, aspirin, etc.);
* Congenital or acquired immunodeficiency; Or receive systemic corticosteroid treatment (any medication route, ≥ 2mg/kg/day) for ≥ 14 days within 3 months prior to enrollment, such as prednisone, inhaled steroids budesonide, fluticasone, etc; Or being using other immunosuppressants such as cyclosporine, tacrolimus, etc. before enrollment;
* Has given immunoglobulin and/or any blood products (except hepatitis B immunoglobulin) within 3 months before enrollment;
* Plan to move before the end of the study visit or leave the local area for a long time during the scheduled study visit;
* Plan to participate or be participating in any other drug clinical research;
* According to the researcher's judgment, there are any other factors that are not suitable for the subjects to participate in the clinical trial.

For booster immunization stage (applicable to the 6-11 month age group) and immune persistence stage (applicable to the 12-23 month age group):

* Subjects in the experimental group aged 6-11 months received any meningococcal vaccine before blood serum collection at 18 months old after completing basic immunization;
* Subjects in the 12-23 month age group were vaccinated with any meningococcal vaccine before completing blood collection at 12 month post-completion of primary immunization schedule;
* After participating in this clinical trial, the subjects are known or suspected to have immunological deficiencies, including being treated with immunosuppressants (such as radiation therapy, chemotherapy, corticosteroids, anti metabolic drugs, cytotoxic drugs, etc.) and HIV infection;
* Subjects in the experimental group aged 6-11 month old were given immunoglobulin and/or any blood products (except hepatitis B immunoglobulin) within 3 months before the booster immunization.
* According to the researcher's judgment, there are any other factors that are not suitable for the subjects to participate in the clinical trial

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2450 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Antibody positive conversion rate | 30 day after primary immunization
  Immunogenicity study of Meningococcal ACYW135 Polysaccharide Conjugate Vaccine as assessed by positive conversion rate (4-fold increase)

CONTACTS AND LOCATIONS:
Overall Officials: Lin Du, Study Chair — Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd
Locations (1):
- Hunan Center for Disease Control and Prevention, Changsha, Hunan, China